CLINICAL TRIAL: NCT04356612
Title: Barriers to Efficient PACU Discharge at a Major Academic Orthopaedic Ambulatory Surgery Center
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-1643
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Achilles Tendon Rupture; Database

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Achilles Tendon Rupture: This is a retrospective chart review to determine the etiologies contributing to prolonged PACU discharge at a major Orthopedic Ambulatory Surgical Center.
  Interventions: Other: Chart Review

INTERVENTIONS:
Other: Chart Review — This is a retrospective chart review to determine the etiologies contributing to prolonged PACU discharge at a major Orthopedic Ambulatory Surgical Center.

SUMMARY:
This is a retrospective chart review to determine the etiologies contributing to prolonged PACU discharge at a major Orthopedic Ambulatory Center

DETAILED DESCRIPTION:
Increasing number of surgeries are now performed at ambulatory surgical centers including orthopaedic procedures. While healthier patients usually undergo non-major orthopaedic procedures using regional anesthesia to facilitate faster discharges, prolonged PACU discharges are frequently encountered necessitating characterization and identification of modifiable variables. This is a retrospective chart review to determine the etiologies contributing to prolonged PACU discharge at a major Orthopedic Ambulatory Center.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years and older) undergoing ambulatory foot and ankle surgery

Exclusion Criteria:

* n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients undergoing ambulatory foot and ankle surgery
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-12-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Time required for discharge | Day of surgery (Day 0) through discharge, average of 6 hours
  This is the length of time that patients stay in the recovery room

SECONDARY OUTCOMES:
Supplemental Analgesics | Day of surgery (Day 0) through discharge, average of 6 hours
  This is the amount of pain medication patients require in the recovery room

CONTACTS AND LOCATIONS:
Overall Officials: Sang Kim, MD, Principal Investigator — Hospital for Special Surgey
Locations (1):
- Hospital for Special Surgery, New York, New York, United States